CLINICAL TRIAL: NCT03897140
Title: Study for Point-of-Care Echocardiography With Assistance Technology
Brief Title: Point-of-Care Echocardiography With Assistance Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Guttas (Industry)
Responsible Party: Sponsor-Investigator, Sara Guttas, Clinical Applications Manager, Caption Health, Inc.
Organization: Caption Health, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EchoGPSPivotal1.0
Record Dates: First submitted 2019-03-23; First posted 2019-04-01 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Patients scheduled for an echocardiogram (Experimental): Patients ≥18 years scheduled for an echocardiographic examination. This is a non-randomized, un-blinded, study in patients with an indication for an echocardiographic examination. Enrolled patients will be stratified into two groups based on known cardiac abnormalities to ensure a sufficient number of patients with cardiac abnormalities and into 3 strata of BMI: normal, overweight and obese.
  Interventions: Diagnostic Test: Diagnostic Test: Limited Echocardiogram

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Limited Echocardiogram — STUDY SOFTWARE non-significant risk (NSR) Bay Labs EchoGPS software interfaced with the Terason uSmart 3200t FDA 510(k)-cleared, commercially available ultrasound EchoGPS software communicates with the ultrasound image formation engine of the 510(k)-cleared Terason uSmart 3200t through an application programming interface (API). EchoGPS will be used to provide visual guidance feedback to users during image acquisition. For this study, RNs will use EchoGPS to perform limited echocardiogram examinations.

SUMMARY:
Establish the effectiveness of the Bay Labs, Inc. EchoGPS software in enabling RNs to acquire echocardiograms. In this study an echocardiogram protocol using the EchoGPS interface with the Terason uSmart 3200t, an FDA 510(k)-cleared, commercially available ultrasound device will be performed. Participants will have two scans, one by a registered nurse (RN) using the Terason uSmart 3200t with EchoGPS (Study Exam) and one by a sonographer using the Reference Device without EchoGPS guidance (Control Exam), under the same protocol. Study is non-significant risk (NSR).

DETAILED DESCRIPTION:
To validate clinical use of Bay Labs, Inc. EchoGPS guidance software by registered nurses (RNs) with no prior scanning experience to acquire limited two-dimensional echocardiograms. In this study an echocardiogram protocol using the EchoGPS interface with the Terason uSmart 3200t, an FDA 510(k)-cleared, commercially available ultrasound device will be performed. Participants will have two scans, one by a registered nurse (RN) using the Terason uSmart 3200t with EchoGPS (Study Exam) and one by a sonographer using the Reference Device without EchoGPS guidance (Control Exam), under the same protocol. Study is non-significant risk (NSR).

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following inclusion criteria to participate in the study:

* Patients scheduled for an echocardiographic examination
* Patients ≥18 years old

Exclusion Criteria:

Patients must NOT meet any of the following exclusion criteria to participate in the trial:

* Unable to lie flat for study
* Patients experiencing a known or suspected acute cardiac event
* Patients with severe chest wall abnormalities
* Patients who have undergone pneumonectomy
* Patients unwilling or unable to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Study-level Assessment | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  The primary endpoints for the study are separate patient-level assessments of whether the patient study is of adequate image quality to make a qualitative visual assessment for a particular clinical parameter (ie., Yes/No). Expert cardiologist readers will independently provide assessments and they will be blinded to the assessments from the other readers as well as whether the images were acquired by an RN or sonographer.
  The Outcome Measure will be reported as the percentage of patient studies for which the panel of cardiologist readers adjudicated as being of sufficient image quality to make a particular clinical assessment.

SECONDARY OUTCOMES:
View-level Assessment | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  The Outcome Measure will be reported as the percentage of patient studies with diagnostic quality clip for a particular Standard View acquired in the study. Expert cardiologist readers will independently provide assessments and they will be blinded to the assessments from the other readers as well as whether the images were acquired by an RN or sonographer.
Inter-User Variability (Primary Clinical Parameters) | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  o Comparison of user variability for primary clinical parameters (measured as the coefficient variation for binary assessment of whether the study is of diagnostic quality to make a particular clinical assessment)
Inter-User Variability (Acquisition Time) | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  o View level acquisition time (minutes and seconds)
Patient-Level Acquisition time | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  o Patient level acquisition time (minutes and seconds)
View-Level Acquisition time | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  o View-level acquisition time (minutes and seconds)
Comparison of study exam and control exam (View-Level Results) | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  o Comparison of View level results measured as percent agreement of images with diagnostic quality
Comparison of study exam and control exam (Patient-Level Results) | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  o Comparison of patient level results measured as percent agreement of patient exams of sufficient quality to make a particular clinical assessment
Comparison of study exam and control exam (Task-Based Assessment) | Up to 2 months from the completion of the study or when all expert cardiologists readers independently complete their assessments
  o Comparison of qualitative assessments from study and control exam to assess whether cardiologists reach a similar decision with study exam images and control exam images

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Narang, MD, Principal Investigator — Northwestern Medicine, Bluhm Cardiovascular Institute
Locations (2):
- United States (2):
  - Northwestern Medicine, Bluhm Cardiovascular Institute, Chicago, Illinois
  - Minneapolis Heart Institute, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will not be made available to other researchers.
Time Frame: N/A - IPD will not be made available to other researchers.
Access Criteria: N/A - IPD will not be made available to other researchers.